CLINICAL TRIAL: NCT07137702
Title: Impact of Erector Spinae Plane Block on Systemic Immune-inflammation Index in Breast-conserving Surgery: A Retrospective Cohort Study
Brief Title: Impact of Erector Spinae Plane Block on Systemic Immune-inflammation Index
Status: Completed | Type: Observational
Sponsor: Taner Abdullah (Other)
Responsible Party: Sponsor-Investigator, Taner Abdullah, MD, Istanbul Saglik Bilimleri University
Organization: Istanbul Saglik Bilimleri University (Other)
Other Study IDs: 2025-225
Record Dates: First submitted 2025-08-16; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Systemic Immune-inflammatory Index; Erector Spinae Plane Block; Breast Conserving Surgery
Keywords: systemic immune-inflammatory index; erector spinae plane block; breast conserving surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ESPB + group: the patients who received erector spinae plane block
  Interventions: Procedure: Erector Spinae Plane Block
- ESPB - group: the patients who didn't receive erector spinae plane block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — A standardized perioperative care management protocol is applied for all breast-conserving surgery procedures in our department. All patients are informed about ESPB and offered its application preoperatively. Patients who accept the procedure receive ESPB (preoperatively, in the sitting position, at the level of ipsilateral T4 vertebra, USG guided, out-of-plane approach) while those who refuse are subjected to routine intravenous analgesia protocols. All blocks were performed by an anesthesiologist experienced in the application of truncal blocks and 20 cc 0.5% bupivacaine (within the safe dose range for all patients to be used according to their weight) are injected and its spread is visualized under USG.
  Groups: ESPB + group

SUMMARY:
The primary objective of the study is to determine whether there is a relationship between postoperative SII and erector spinae plane block application. If data emerges indicating a more suppressed inflammatory response in patients undergoing block, widespread use of this block in the specified patient group would reflect the clinical significance of the study.

The searches did not uncover any studies investigating the effects of trunk blocks, such as erector spinae plane block, on postoperative systemic inflammatory response, indicating that this study could make a significant contribution to the literature.

DETAILED DESCRIPTION:
Because the study will be conducted retrospectively, it carries no potential risks.

If it can be demonstrated that blocking has a suppressive effect on the inflammatory response, the main expected benefit of the study is its widespread use to improve postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria: ASA score ≤ 3, breast-conversing surgery, age > 18 -

Exclusion Criteria: ASA score > 3, reoperation, surgical wound infection, chemotherapy in less than 2 weeks, bening lesions

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women who have undergone breast-conserving surgery for malignant causes
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
systemic immune-inflammation index | 7 days after surgery
  Platelet count × Neutrophil count / Lymphocyte count

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Cam ve Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No